Version 1.0, 08-SEP-2022

**Protocol Number: Careseng 1370-01** 

A Phase I Dose-Escalation Study in Healthy Volunteers to Evaluate the Safety and Tolerability Profiles of Careseng 1370

Protocol version: 5.0, 18SEP2020

Sponsor:

Version 1.0, 08-SEP-2022 Protocol No.: Careseng 1370-01 

A2 Healthcare Taiwan Co.

## **Statistical Analysis Plan: Mock-up Tables and Figures** Careseng 1370 for Healthy Volunteers

#### **Table of Contents**

| Statistical | Analysis Plan: Mock-up Tables and Figures | 1 |
|-------------|-----------------------------------------------|----|
| Table of C | ontents | 2 |
| 1 Stati | stical Changes from Study Protocol | 3 |
| 1.1 | Visit Adjustment | |
| 1.2 | Analysis Populations | |
| 1.3 | Treatment Compliance | |
| 1.4 | Pharmacokinetic Analysis | |
| 3 Prote | ocol Versions and Protocol Amendments | 4 |
| 4 Mocl | ι-up Tables and Figures | 5 |
| | s and Abbreviations: | |
| | LES and FIGURES | |
| 14.1 | DEMOGRAPHIC DATA AND BASELINE CHARACTERISTICS | |
| 14.1. | | |
| 14.1. | | 9 |
| 14.1. | | 10 |
| 14.1. | · | |
| 14.1. | ,,,,,,,,,, | |
| 14.1. | | |
| 14.2 | EFFICACY DATA | 11 |
| 14.3 | SAFETY DATA | 12 |
| 14.3. | | |
| 14.3. | 2 Laboratory Examination – Hematology | 16 |
| 14.3. | B Laboratory Examination – Biochemistry | 16 |
| 14.3. | | |
| 14.3. | 5 Laboratory Examination – Immunology | 16 |
| 14.3. | 6 Physical Examination | 19 |
| 14.3. | 7 Vital Signs and Body Weight | 19 |
| 14.3. | 3 12-Lead Electrocardiogram (EKG) | 20 |

Careseng 1370 for Healthy Volunteers

#### 1 Statistical Changes from Study Protocol

The statistical analysis methods will follow study protocol version 5.0, (18SEP2020), exceptions and clarifications are described below:

#### 1.1 Visit Adjustment

Visit 11 is final visit or early withdrawal visit, refer to 14.3 for detail of visit adjustment

#### 1.2 Analysis Populations

According to the protocol, only Intent-to-treat (ITT) population was defined for analyses of primary and secondary endpoints.

Section 10.2.1 Analysis Population: Intent-to-treat (ITT) population:

- Volunteers receive any Careseng 1370

For maximal tolerated dose (MTD) determination, a MTD-Evaluable Population is defined as below according to protocol section 3.1 "Volunteers Enrollment" on DLT analysis.

MTD-Evaluable Population:

- 1. A subset of ITT population
- 2. Experiences DLT OR completes DLT observation period with at least 80% of study drug compliance and has exposed to Careseng 1370 for at least 4 days (level A, B, and C), OR completes DLT observation period with 100% of study drug compliance (level D).

#### 1.3 Treatment Compliance

Treatment compliance is defined as below in protocol section 5.6:

| Volunteer's compliance will be assessed by the following formula: | |
|-------------------------------------------------------------------|----------|
| # of sachets of study drug actually administered | - × 100% |
| Total # of sachets of study drug assigned at that level | - × 100% |

The parameters of compliance calculation are not well-defined in the protocol. The formula to derive treatment compliance and relevant parameters are adjusted as below:

```
Treatment Compliance = # of sachets of study drug actually administered

Dose Level [Sachet/Day] × Treatment Duration × 100%

[Days]
```

• Treatment Duration [Days] = the last dosing date - the first dosing date + 1.

## 1.4 Pharmacokinetic Analysis

Pharmacokinetic parameters will be analyzed by Mithra Biotechnology Inc. All pharmacokinetic parameters data will be provided to sponsor directly, no data handling, data listing nor statistical analysis on such data will be done by A2 Healthcare.

- 2.2 Endpoints
  - 2.2.2 Secondary endpoints
    - 2 Pharmacokinetic parameters of marker ingredient in Careseng 1370, 20(S)-protopanaxadiol (PPD) and its metabolites



Careseng 1370 for Healthy Volunteers

#### 3 Protocol Versions and Protocol Amendments

The first subject was enrolled on 14AUG2020, and the last subject is expected to be dismissed on MAR2022. Amendments relevant to important statistical-related changes are summarized in table below, and Table/Figure/Listing programming will be based on the latest version of protocol.

| Summary of important statistical-related changes for protocol version V4.0 |
|----------------------------------------------------------------------------|
| Additional time points for PK blood sampling for Dose level B and C |

Summary of important statistical-related changes for protocol version V5.0

Addition of 1 lower dose cohort (level D), and the corresponding information

Version 1.0, 08-SEP-2022 Protocol No.: Careseng 1370-01



Careseng 1370 for Healthy Volunteers

#### 4 Mock-up Tables and Figures

The Mock-up "TABLES and FIGURES" is planned according to ICH E3, in which relevant CSR section is 14. The words shadowed below are to be adjusted or repeated upon real data, or just for notification.

Columns {Label, Dose Level} will be included in the table with the analyzed population specified. In the mock table below, only the Label with one dose level column were presented to show the descriptive/inferential statistics to be displayed in the final tabulation.

Version 1.0, 08-SEP-2022 Protocol No.: Careseng 1370-01 



Careseng 1370 for Healthy Volunteers

#### **Instructions and Abbreviations:**

(1) Site ID [C]:

| Site ID | Full Name |
|---------|-------------------------------------------|
| 1 | Taipei Medical University Hospital (TMUH) |

#### (2) Dose Level:

- A (1 sachet/day): Careseng 1370 1 sachet before breakfast for consecutive 5 days
- B (2 sachets/day): Careseng 1370 1 sachet before breakfast and 1 sachet before lunch for consecutive 5 days
- C (3 sachets/day): Careseng 1370 1 sachet before breakfast and 2 sachets before lunch for consecutive 5 days
- D (1 sachet/day): Careseng 1370 1 sachet before breakfast on 1st, 3rd and 5th days (modified cohort)

#### (3) Population

- Intention-to-Treat (ITT) Population:
  - Volunteers receive any Careseng 1370
- Maximum Tolerated Dose (MTD)-Evaluable Population:
  - 1. A subset of ITT population
  - 2. Experiences DLT OR with at least 80% of study drug compliance and has exposed to Careseng 1370 for at least 4 days

(4) For Visit Name (in Tables and Figures) and Visit Code (in Subject Data Listing):

| Visit No. | Visit Description | Visit Day | Visit Name | Visit Code |
|---|---|---|---|---|
| 1 | Visit 1 Screening Visit | <b>-14</b> ∼ <b>-1</b> | Visit 1 (Screening) | V01 |
| 2 | Visit 2 Hospitalization: Day -1 to Day 1 | 1 | Visit 2 (Day 1) | V02D01 |
| 3 | Visit 3 Discharge: Day 2 | 2 | Visit 3 (Day 2) | V03D02 |
| 4 | Visit 4: Day 3 | 3 | Visit 4 (Day 3) | V04D03 |
| 5 | Visit 5: Day 4 | 4 | Visit 5 (Day 4) | V05D04 |
| 6 | Visit 6 Hospitalization: Day 4 to Day 5 | 5 | Visit 6 (Day 5) | V06D05 |
| 7 | Visit 7 Discharge: Day 6 (24±2 hrs post-last dose) | 6 | Visit 7 (Day 6) | V07D06 |
| 8 | Visit 8 Follow-up Visit: Day 7 (48±2 hrs post-last dose) | 7 | Visit 8 (Day 7) | V08D07 |
| 9 | Visit 9 Follow-up Visit: Day 8 (72±2 hrs post-last dose) | 8 | Visit 9 (Day 8) | V09D08 |
| 10 | Visit 10 Follow-up Visit: Day 12±2 | 10 ~ 14 | Visit 10 (Day 12) | V10D12 |
| 11 | Visit 11 Final Visit (Day 22±2, within 3 days after withdrawal) | 22 | Visit 11 (Day 22) | V11D22 |
| - | Unscheduled Visit | - | - | V□□.□ |

(5) Full term for 'Protocol Deviation Code':

| Code | Full Term |
|---|---|
| <to added="" be="" data="" final="" in="" real="" tabulation="" upon=""></to> | |

(6) For clinical relevance

CS: abnormal and clinically significant LLN: lower limit of normal range NCS: abnormal but not clinically significant ULN: upper limit of normal range

(7) For Transition of Clinical Relevance

Relieved CS (Medical History or Adverse Event) at baseline to Normal / NCS at

visit.

Unchanged Including Normal at baseline to NCS at visit, NCS at baseline to Normal

at visit.

Worsened (Medical History) Normal / NCS at baseline to CS (Medical History) at visit

Worsened (Adverse Event) Normal / NCS / CS (Medical History) at baseline to CS (Adverse Event)

at visit

Version 1.0, 08-SEP-2022 Confidential
Protocol No.: Careseng 1370-01  A2 Healthcare Taiwan Co.



Careseng 1370 for Healthy Volunteers

(8) Abbreviations of statistics

N: number of non-missing values Missing: number of missing values

Mean: mean of values

SD: standard deviation of values Q1: 25% quartile of values Q3: 75% quartile of values

Median: median of values

IQR: inter-quartile-range (IQR=Q3-Q1)

Min: minimum of values Max: maximum of values CI: confidence interval

Version 1.0, 08-SEP-2022 C Protocol No.: Careseng 1370-01 P



Careseng 1370 for Healthy Volunteers

#### 14 TABLES AND FIGURES

- The texts in shaded Italic are for programming note.
- Column of Study Site includes {Site 1: TMUH}
- Column of Dose Level includes {A (1 sachet/day), B (2 sachets/day), C (3 sachets/day), D (1 sachet/day), Total} as appropriate
- Description in <...> will be presented according to data values.

#### 14.1 DEMOGRAPHIC DATA AND BASELINE CHARACTERISTICS

## 14.1.1 Screen Failures and Subject Disposition by Study Site

| Characteristics | Study Site |
|--------------------------------------------------|---------------|
| .All Screened Subjects | ****** |
| n | XXX |
| Eligible Subjects | XXX (XXX.X%) |
| Screening Failures | XXX (XXX.X%) |
| <screen 1="" failure="" reason=""></screen> | XXX (XXX.X%) |
| <screen 2="" failure="" reason=""></screen> | XXX (XXX.X%) |
| <screen 3="" failure="" reason=""></screen> | XXX (XXX.X%) |
| | XXX (XXX.X%) |
| .Population of Eligible Subjects | |
| n | XXX |
| ITT | XXX (XXX.X%) |
| MTD-Evaluable | XXX (XXX.X%) |
| Non-MTD-Evaluable | XXX (XXX.X%) |
| <reason 1=""></reason> | XXX (XXX.X%) |
| <reason 2=""></reason> | XXX (XXX.X%) |
| | XXX (XXX.X%) |
| Non-ITT | XXX (XXX.X%) |
| Daga Lavel of Elicikla Cukiasta | |
| .Dose Level of Eligible Subjects | XXX |
| A (1 sachet/day) | |
| | XXX (XXX.X%) |
| B (2 sachets/day) | XXX (XXX.X%) |
| C (3 sachets/day) | XXX (XXX.X%) |
| D (1 sachet/day) | XXX (XXX.X%) |
| . Protocol Deviation of Eligible Subjects | |
| n | XXX |
| Major Protocol Deviation | XXX (XXX.X%) |
| <protocol 1="" deviation=""></protocol> | XXX (XXX.X%) |
| <protocol 2="" deviation=""></protocol> | XXX (XXX.X%) |
| <br>Minor Protocol Deviction | VVV (VVV V0/) |
| Minor Protocol Deviation | XXX (XXX.X%) |
| <pre><pre><pre><pre>&lt;</pre></pre></pre></pre> | XXX (XXX.X%) |
| <protocol 2="" deviation=""></protocol> | XXX (XXX.X%) |

ITT: Intent-to-Treat population, MTD-Evaluable: Maximum Tolerated Dose-Evaluable Population (subset of ITT)



Careseng 1370 for Healthy Volunteers

# 14.1.2 Study Visits, Study Termination, Subject Disposition and Protocol Deviation

| Population: Intent-to-Treat Population | |
|---|---|
| Characteristics | Dose Level |
| . Study Termination | |
| n | XXX |
| Study Completed | XXX (XXX.X%) |
| Study Not Completed | XXX (XXX.X%) |
| Withdrew consent | XXX (XXX.X%) |
| Protocol issue | XXX (XXX.X%) |
| ••• | XXX (XXX.X%) |
| . Study Duration [days] | |
| n (Missing) | XXX |
| Mean (SD) | XXX (XXX) |
| Median (IQR) | XXX (XXX) |
| Q1~Q3 | XXX~XXX |
| Min~Max | XXX~XXX |
| .Population | ***** |
| n<br>NATE E 1 11 | XXX |
| MTD-Evaluable | XXX (XXX.X%) |
| Non-MTD-Evaluable | XXX (XXX.X%) |
| <reason 1=""></reason> | XXX (XXX.X%) |
| <reason 2=""></reason> | XXX (XXX.X%) |
| | XXX (XXX.X%) |
| .Protocol Deviation | |
| n | XXX |
| Major Protocol Deviation | XXX (XXX.X%) |
| <protocol 1="" deviation=""></protocol> | XXX (XXX.X%) |
| <protocol 2="" deviation=""></protocol> | XXX (XXX.X%) |
| Minor Protocol Deviation | XXX (XXX.X%) |
| <protocol 1="" deviation=""></protocol> | XXX (XXX.X%) |
| <protocol 2="" deviation=""></protocol> | XXX (XXX.X%) |
| . Study Visits Completed, Adjusted Visits Completed | |
| N | XXX |
| Visit 1 (Screening) | XXX (XXX.X%) |
| Visit 2 (Day 1) | XXX (XXX.X%) |
| Visit 3 (Day 2) | XXX (XXX.X%) |
| Visit 4 (Day 3)<br>Visit 5 (Day 4) | XXX (XXX.X%)<br>XXX (XXX.X%) |
| Visit 5 (Day 4)<br>Visit 6 (Day 5) | XXX (XXX.X%) $XXX (XXX.X%)$ |
| Visit 7 (Day 6) | XXX (XXX.X%) |
| Visit 8 (Day 7) | XXX (XXX.X%) |
| Visit 9 (Day 8) | XXX (XXX.X%) |
| Visit 10 (Day 12) | XXX (XXX.X%) |
| Visit 11 (Day 22) | XXX (XXX.X%) |

Study Duration [days] = Date of Termination - Visit 1, or alternatively as the last visit date - Visit 1 Adjusted Visits Completed: Visits except visit 8 and visit 9 not in its visit window are shifted to corresponding scheduled visits



Careseng 1370 for Healthy Volunteers

## 14.1.3 Demographic Data

| Characteristics | Dose Level |
|------------------------------------------------------------|--------------|
| . Study Sites | |
| n (Missing) | XXX (XXX) |
| Site 1: TMUH | XXX (XXX.X%) |
| . Variable, including Age [Y/O], Baseline Body Weight [kg] | , Height |
| [cm], BMI [kg/m^2] | |
| n (Missing) | XXX (XXX) |
| Mean (SD) | XXX (XXX) |
| Median (IQR) | XXX (XXX) |
| Q1~Q3 | XXX~XXX |
| Min~Max | XXX~XXX |
| . Gender | |
| n (Missing) | XXX (XXX) |
| Male | XXX (XXX.X%) |
| Female | XXX (XXX.X%) |
| . Race (multiple selection) | |
| n (Missing) | XXX (XXX) |
| Black or African American | XXX (XXX.X%) |
| American Indian or Alaska Native | XXX (XXX.X%) |
| Asian | XXX (XXX.X%) |
| Native Hawaiian or Other Pacific Islander | XXX (XXX.X%) |
| White | XXX (XXX.X%) |
| Not Reported | XXX (XXX.X%) |
| Unknown | XXX (XXX.X%) |

Age [Y/O] = int((date of informed consent - date of birth)/365.25)

BMI [kg/m $^2$ ]= Weight [kg] / (Height [cm]) $^2 * 10000$ 

Baseline is Visit 2 or alternatively as Visit 1 if Visit 2 data is not available

# 14.1.4 General Medical History, Concurrent Disease/Status and Chest X-Ray

Population: Intent-to-Treat Population

| Characteristics | Dose Level |
|------------------------------|--------------|
| .General Medical History | |
| n | XXX |
| At least one below | XXX (XXX.X%) |
| <body 1="" system=""></body> | XXX (XXX.X%) |
| <body 2="" system=""></body> | XXX (XXX.X%) |
| <body 3="" system=""></body> | XXX (XXX.X%) |
| <body 4="" system=""></body> | XXX (XXX.X%) |
| . Current Condition | |
| n | XXX |
| At least one below | XXX (XXX.X%) |
| <body 1="" system=""></body> | XXX (XXX.X%) |
| <body 2="" system=""></body> | XXX (XXX.X%) |
| <body 3="" system=""></body> | XXX (XXX.X%) |
| <body 4="" system=""></body> | XXX (XXX.X%) |
| *** | ••• |

Version 1.0, 08-SEP-2022 Protocol No.: Careseng 1370-01



Careseng 1370 for Healthy Volunteers

| Characteristics | Dose Level |
|----------------------|-------------|
| n (Missing) | XXX (XXX) |
| Normal | XXX (XX.X%) |
| NCS | XXX (XX.X%) |
| CS (Medical History) | XXX (XX.X%) |
| CS (Adverse Event) | XXX (XX.X%) |
| Not Interpretable | XXX (XX.X%) |

Current condition lists the medical histories that are ongoing or with end date  $\geq$  date of visit 2

#### 14.1.5 Prohibited Medications, Treatments, Procedures and Foods

For Prohibited Medications, categories are Surgery, Herbal Medications, Herbal Supplements, Herbal Medicinal Food, Other. For Prohibited Foods, refer to CRF for the categories.

Population: Intent-to-Treat Population

| _ 1 | |
|--------------------------------------------------|--------------|
| Characteristics | Dose Level |
| . Prohibited Medications, Treatments, Procedures | |
| . Prohibited Foods | |
| n (Missing) | XXX (XXX) |
| At least one below | XXX (XXX.X%) |
| <category 1=""></category> | XXX (XXX.X%) |
| <category 2=""></category> | XXX (XXX.X%) |
| <category 3=""></category> | XXX (XXX.X%) |
| <category 4=""></category> | XXX (XXX.X%) |
| | ••• |

#### 14.1.6 Study Drug Administration, Compliance and Exposure

Population: Intent-to-Treat Population

| Characteristics | Dose Level |
|-------------------------------------|--------------|
| .Total IP Administration [sachets], | |
| Treatment Duration [days] | |
| Treatment Compliance [%], | |
| Mean Daily Dose [sachet/day] | |
| n (Missing) | XXX |
| Mean (SD) | XXX (XXX) |
| Median (IQR) | XXX (XXX) |
| Q1~Q3 | XXX~XXX |
| Min~Max | XXX~XXX |
| . Treatment Compliance | |
| n (Missing) | XXX (XXX) |
| <60% | XXX (XXX.X%) |
| 60 ~ <80% | XXX (XXX.X%) |
| 80 ~ < 100% | XXX (XXX.X%) |
| 100 ~ <120% | XXX (XXX.X%) |
| ≥120% | XXX (XXX.X%) |

- Treatment Duration [days] = the last dosing date the first dosing date + 1.
- Treatment Compliance [%] = Total IP Administration [sachets] / Dose Level [sachet/day] / Treatment Duration [days] \* 100%
- Mean Daily Dose [sachet/day] = Total IP Administration [sachets] / Treatment Duration [days]

#### 14.2 EFFICACY DATA

N/A



Careseng 1370 for Healthy Volunteers

#### 14.3 SAFETY DATA

Visit 11 is final visit or early withdrawal visit.

Safety data below except for visit 8 and visit 9 not in its visit window will be shifted to corresponding scheduled visit for analysis as in table below. If there is any data shifting, visit name will be presented as 'Adjusted Visit' for the visits reallocated to its original scheduled visit or the next visit after preceding scheduled visit.

| Adjusted Visit | Laboratory<br>Assessment† | Physical<br>Examination | Body Weight | Vital Signs | 12-Lead<br>Electrocardiogram |
|---|---|---|---|---|---|
| Baseline | N Baseline is Visit 1 (Screening), no need to present statistics for Baseline additionally | N. | Y Baseline is Day 1, or alternatively as Visit 1 if Day 1 data are not available. | Y Baseline is Day 1 Pre-dose, or alternatively as Visit 1 if Day 1 Pre-dose data are not available. | Y Baseline is Day 1 Predose, or alternatively as Visit 1 if Day 1 Predose data are not available. |
| • Visit 1 | Y | Y | Y | Y | Y |
| • Visit 2 (Day 1) | Y<br>(8 hours post-first<br>dose) | Y<br>(Pre-dose),<br>(8 hours post-<br>first dose) | Y | Y (Pre-dose), (1 hour post-first dose), (4 hours post-first dose), (8 hours post-first dose) | Y (Pre-dose), (1 hour post-first dose), (4 hours post-first dose), (8 hours post-first dose), (12 hours post-first dose) |
| • Visit 3 (Day 2) | Y | Y | Y | Y | Y<br>(Pre-dose),<br>(1 hour post-first dosing<br>post-first dosing) |
| • Visit 4 (Day 3) | Y | Y | Y | Y | Y (Pre-dose), (1 hour post-first dosing) |
| • Visit 5 (Day 4) | Y | Y | Y | Y | Y (Pre-dose),<br>(1 hour post-first dosing) |
| • Visit 6 (Day 5) | Y<br>(Pre-dose),<br>(4 hours post dosing) | Y<br>(Pre-dose),<br>(4 hours post<br>dosing) | Y | Y<br>(Pre-dose),<br>(4 hours post dosing) | Y (Pre-dose), (1 hour post-first dose), (4 hours post-first dose), (8 hours post-first dose), (12 hours post-first dose) |
| • Visit 7 (Day 6) | Y | Y | Y | Y | Y |
| • Visit 8 (Day 7) | N | N | N | N | N |
| • Visit 9 (Day 8) | N | N | N | N | N |
| • Visit 10 (Day 12) | Y | Y | Y | Y | Y |
| • Visit 11 (Day 22) | Y | Y | Y | Y | Y |

Y denotes that the Visit is performed in the corresponding tables.

N denotes that the Visit is not performed in the corresponding tables.

<sup>†</sup> Visit 1, 3, 7, 11 only for immunology



Careseng 1370 for Healthy Volunteers

#### 14.3.1 Treatment Emergent Adverse Event – Subject Based Analyses

For 14.3.1.4, population will include ITT and MTD-Evaluable population.

#### 14.3.1.1 Treatment Emergent AE - Summary

Population: Intent-to-Treat Population / MTD-Evaluable Population

| Characteristics [Event#:Subj#] | Treatment |
|---|---|
| Repeat Population: Intent-to-Treat Population, MTD- | Evaluable Population |
| n | XXX |
| Subjects with AE | XXX : XXX (XXX.X%) |
| Subjects with Treatment-Related AE | XXX : XXX (XXX.X%) |
| Subjects with DLT | XXX : XXX (XXX.X%) |
| Subjects with Grade ≥3 AE | XXX : XXX (XXX.X%) |
| Subjects with Grade ≥3 Treatment-Related AE | XXX : XXX (XXX.X%) |
| Subjects with AE Leading to Action Taken | XXX : XXX (XXX.X%) |
| Subjects with AE Leading to Drug withdrawn | XXX : XXX (XXX.X%) |
| Subjects with SAE | XXX : XXX (XXX.X%) |
| Subjects with Death SAE | XXX : XXX (XXX.X%) |
| Subjects with SUSAR | XXX : XXX (XXX.X%) |
| Subjects with Death SUSAR | XXX: XXX (XXX.X%) |

Subject with multiple events are counted as one incidence.

Treatment-Related is defined as Definitely Related, Probable Related, or Possibly Related

Programmer's Notes:

Repeat Population only when the two populations are not identical

#### 14.3.1.2 Treatment Emergent AE - Subjects with AE

#### 14.3.1.3 Treatment Emergent AE - Subjects with Treatment-Related AE

#### 14.3.1.4 Treatment Emergent AE – Subjects with DLT

[For 14.3.1.2-3] Population: Intent-to-Treat Population

[For 14.3.1.4] Population: Intent-to-Treat Population / MTD-Evaluable Population

| Characteristics [Event#:Subj#] | Dose Level |
|---|---|
| Repeat Population: Intent-to-Treat Population, MT | TD-Evaluable Population (Applied for |
| 14.3.1.4) | |
| . By MedDRA SOC and Preferred Term | |
| n | XXX |
| At least one below | XXX : XXX (XXX.X%) |
| <meddra 1="" body="" system=""></meddra> | XXX : XXX (XXX.X%) |
| <meddra 1="" preferred="" term=""></meddra> | XXX : XXX (XXX.X%) |
| <meddra 2="" preferred="" term=""></meddra> | XXX : XXX (XXX.X%) |
| <meddra 3="" preferred="" term=""></meddra> | XXX : XXX (XXX.X%) |
| | XXX : XXX (XXX.X%) |
| <meddra 2="" body="" system=""></meddra> | XXX : XXX (XXX.X%) |
| <meddra 1="" preferred="" term=""></meddra> | XXX : XXX (XXX.X%) |
| <meddra 2="" preferred="" term=""></meddra> | XXX : XXX (XXX.X%) |
| <meddra 3="" preferred="" term=""></meddra> | XXX : XXX (XXX.X%) |

For each MedDRA (version 23.0) SOC or Preferred Term, Subject with multiple events are counted as one incidence

[For 14.3.1.3] Treatment-Related is defined as Definitely Related, Probable Related, or Possibly Related

Programmer's Notes:

Repeat Population only when the two populations are not identical

Sorted in descending order of Subject No, Event No. of Total column by MedDRA Body System first, and then MedDRA Preferred Term.

Version 1.0, 08-SEP-2022 Confidential
Protocol No.: Careseng 1370-01 



Careseng 1370 for Healthy Volunteers

#### 14.3.1.5 Treatment Emergent AE - Subjects with Grade ≥3 AE

#### 14.3.1.6 Treatment Emergent AE - Subjects with Grade ≥3 Treatment-Related AE

Population: Intent-to-Treat Population

| Characteristics [Event#:Subj#] | Dose Level |
|----------------------------------------------------|--------------------|
| . By Severity Grade, MedDRA SOC and Preferred Term | |
| n | XXX |
| At least one below | XXX: XXX (XXX.X%) |
| Grade ≥3, Grade 4, Grade 5 | XXX: XXX (XXX.X%) |
| <meddra 1="" body="" system=""></meddra> | XXX : XXX (XXX.X%) |
| <meddra 1="" preferred="" term=""></meddra> | XXX : XXX (XXX.X%) |
| <meddra 2="" preferred="" term=""></meddra> | XXX : XXX (XXX.X%) |
| <meddra 3="" preferred="" term=""></meddra> | XXX: XXX (XXX.X%) |
| | XXX: XXX (XXX.X%) |
| <meddra 2="" body="" system=""></meddra> | XXX: XXX (XXX.X%) |
| <meddra 1="" preferred="" term=""></meddra> | XXX : XXX (XXX.X%) |
| <meddra 2="" preferred="" term=""></meddra> | XXX : XXX (XXX.X%) |
| <meddra 3="" preferred="" term=""></meddra> | XXX:XXX(XXX.X%) |

[For 14.3.1.6] Treatment Related is defined as Definitely Related, Probable Related, or Possibly Related

Programmer's Notes:

Sorted in descending order of Subject No, Event No. of Total column by MedDRA Body System first, and then MedDRA Preferred Term for each Grade Level

#### 14.3.1.7 Treatment Emergent AE - Subjects with AE Leading to Action Taken

Population: Intent-to-Treat Population

| r opulation. Intent to Treat r opulation | |
|--------------------------------------------------|--------------------|
| Characteristics [Event#:Subj#] | Dose Level |
| . By Action Taken, MedDRA SOC and Preferred Term | |
| n | XXX |
| At least one below | XXX: XXX (XXX.X%) |
| Drug interrupted, Drug withdrawn | XXX:XXX(XXX.X%) |
| <meddra 1="" body="" system=""></meddra> | XXX : XXX (XXX.X%) |
| <meddra 1="" preferred="" term=""></meddra> | XXX : XXX (XXX.X%) |
| <meddra 2="" preferred="" term=""></meddra> | XXX : XXX (XXX.X%) |
| <meddra 3="" preferred="" term=""></meddra> | XXX: XXX (XXX.X%) |
| <meddra 2="" body="" system=""></meddra> | XXX : XXX (XXX.X%) |
| <meddra 1="" preferred="" term=""></meddra> | XXX : XXX (XXX.X%) |
| <meddra 2="" preferred="" term=""></meddra> | XXX : XXX (XXX.X%) |
| <meddra 3="" preferred="" term=""></meddra> | XXX : XXX (XXX.X%) |

Programmer's Notes:

Sorted in descending order of Subject No, Event No. of Total column by Action Taken first, then MedDRA Body System, and then MedDRA Preferred Term

Version 1.0, 08-SEP-2022 Protocol No.: Careseng 1370-01



Careseng 1370 for Healthy Volunteers

#### 14.3.1.8 Treatment Emergent AE – Subjects with SAE

#### 14.3.1.9 Treatment Emergent AE – Subjects with SUSAR

SUSAR: Suspected Unexpected Serious Adverse Reaction (Unexpected **Treatment Related SAE)** 

Population: Intent-to-Treat Population

| Characteristics [Event#:Subj#] | Dose Level |
|--------------------------------------------------|--------------------|
| . By SAE Criteria, MedDRA SOC and Preferred Term | |
| n | XXX |
| At least one below | XXX: XXX (XXX.X%) |
| <sae criterion=""></sae> | XXX : XXX (XXX.X%) |
| <meddra 1="" body="" system=""></meddra> | |
| <meddra 1="" preferred="" term=""></meddra> | XXX : XXX (XXX.X%) |
| <meddra 2="" preferred="" term=""></meddra> | XXX: XXX (XXX.X%) |
| <meddra 3="" preferred="" term=""></meddra> | XXX: XXX (XXX.X%) |
| | XXX : XXX (XXX.X%) |
| <meddra 2="" body="" system=""></meddra> | |
| <meddra 1="" preferred="" term=""></meddra> | XXX : XXX (XXX.X%) |
| <meddra 2="" preferred="" term=""></meddra> | XXX : XXX (XXX.X%) |
| <meddra 3="" preferred="" term=""></meddra> | XXX: XXX (XXX.X%) |
| | XXX:XXX(XXX.X%) |

SAE Criteria 'F/L/H' and 'F/L' will be counted as 'F' only, and 'L/H' as 'L', where F=Fatal (Death), L=Life threatening, H=Require hospitalization or prolongation of existing hospitalization.

Programmer's Notes:

SAE Criterion: {Any SAE Criterion, Requires or Prolongs Hospitalization, death, ...}

Sorted in descending order of Subject No, Event No. of Total column by SAE Criterion, MedDRA Body System, and

MedDRA Preferred Term



Careseng 1370 for Healthy Volunteers

#### 14.3.2 Laboratory Examination – Hematology

- 14.3.2.1 Hematology < Hematology Item 1 and Unit>
- 14.3.2.2 Hematology < Hematology Item 2 and Unit>
- 14.3.2.3 Hematology < Hematology Item 3 and Unit>
- 14.3.2.4 ...

#### 14.3.3 Laboratory Examination – Biochemistry

- 14.3.3.1 Biochemistry < Biochemistry Item 1 and Unit>
- 14.3.3.2 Biochemistry < Biochemistry Item 2 and Unit>
- 14.3.3.3 Biochemistry < Biochemistry Item 3 and Unit>
- 14.3.3.4 ...

#### 14.3.4 Laboratory Examination – Urinalysis

- **14.3.4.1** Urinalysis pH
- 14.3.4.2 Urinalysis Protein <Unit>
- 14.3.4.3 Urinalysis RBC <Unit>
- 14.3.4.4 Urinalysis WBC <Unit>
- 14.3.4.5 Urinalysis Casts <Unit>

Data '<a', '\secar', '\secar', '\secar' will be estimated as 'a' for analysis.

#### 14.3.5 Laboratory Examination – Immunology

- 14.3.5.1 Immunology CD3 <Unit>
- 14.3.5.2 Immunology CD4 <Unit>
- 14.3.5.3 Immunology CD8 < Unit>
- 14.3.5.4 **Immunology CD16 < Unit >**
- 14.3.5.5 **Immunology CD19 < Unit >**

Version 1.0, 08-SEP-2022 Protocol No.: Careseng 1370-01



Careseng 1370 for Healthy Volunteers

#### <For continuous Laboratory Examination >

Population: Intent-to-Treat Population

| opulation: Intent-to-Treat I opulation | |
|-------------------------------------------------------|-------------|
| Characteristics | Dose Level |
| . (Adjusted) Visits, see visit table below 14.3 | |
| n (Missing) | XXX (XXX) |
| Mean (SD) | XXX (XXX) |
| Median (IQR) | XXX (XXX) |
| Q1~Q3 | XXX~XXX |
| Min~Max | XXX~XXX |
| n (Missing) | XXX (XXX) |
| Normal | XXX (XX.X%) |
| NCS | XXX (XX.X%) |
| CS (Medical History) | XXX (XX.X%) |
| CS (Adverse Event) | XXX (XX.X%) |
| . (Adjusted) Visits - Baseline, see visit table below | |
| n (Missing) | XXX (XXX) |
| Mean (SD) | XXX (XXX) |
| Median (IQR) | XXX (XXX) |
| Q1~Q3 | XXX~XXX |
| Min~Max | XXX~XXX |
| 95% CI (WI) | XXX~XXXwt |
| . Baseline to (Adjusted) Visits, see visit table belo | pw 14.3 |
| n (Missing) | XXX (XXX) |
| Relieved | XXX (XX.X%) |
| Unchanged | XXX (XX.X%) |
| Worsened (Medical History) | XXX (XX.X%) |
| Worsened (Adverse Event) | XXX (XX.X%) |

- For CI (WI, within group), t denotes by using one sample t-test, w denotes CI of median (determined by Shapiro-Wilk normality test)
- Refer to [Instructions and Abbreviations] of title pages for Transition of Clinical Relevance

Programmer's Notes:

Present 'Baseline' as Visit 1 (Screening).



Careseng 1370 for Healthy Volunteers

# **For categorical urinalysis data>**Population: Intent-to-Treat Population

| Population: Intent-to-Treat Population | |
|------------------------------------------------------|-------------|
| Characteristics | Dose Level |
| . (Adjusted) Visits, see visit table below 14.3 | |
| n (Missing) | XXX (XXX) |
| <value 1=""></value> | XXX (XX.X%) |
| <value 2=""></value> | XXX (XX.X%) |
| <value 3=""></value> | XXX (XX.X%) |
| n (Missing) | XXX (XXX) |
| Normal | XXX (XX.X%) |
| NCS | XXX (XX.X%) |
| CS (Medical History) | XXX (XX.X%) |
| CS (Adverse Event) | XXX (XX.X%) |
| Baseline to (Adjusted) Visits, see visit table below | 14.3 |
| n (Missing) | XXX (XXX) |
| <value 1=""></value> | XXX (XX.X%) |
| <value 2=""></value> | XXX (XX.X%) |
| <value 3=""></value> | XXX (XX.X%) |
| Baseline to (Adjusted) Visits, see visit table below | 14.3 |
| n (Missing) | XXX (XXX) |
| Relieved | XXX (XX.X%) |
| Unchanged | XXX (XX.X%) |
| Worsened (Medical History) | XXX (XX.X%) |
| Worsened (Adverse Event) | XXX (XX.X%) |
| , | , |

Refer to [Instructions and Abbreviations] of title pages for Transition of Clinical Relevance

Programmer's Notes:

Present 'Baseline' as Visit 1 (Screening).



Careseng 1370 for Healthy Volunteers

#### 14.3.6 Physical Examination

#### 14.3.6.1 Physical Examination – All Abnormalities

Population: Intent-to-Treat Population

| Characteristics | Dose Level | _ |
|-------------------------------------------------|--------------|---|
| . (Adjusted) Visits, see visit table below 14.3 | | |
| n (Missing) | XXX (XXX) | |
| At least one below | XXX (XXX.X%) | |
| <body 1="" system=""></body> | XXX (XXX.X%) | |
| CS (Medical History) | XXX (XXX.X%) | |
| CS (Adverse Event) | XXX (XXX.X%) | |
| <body 2="" system=""></body> | XXX (XXX.X%) | |
| CS (Medical History) | XXX (XXX.X%) | |
| CS (Adverse Event) | XXX (XXX.X%) | |
| <body 3="" system=""></body> | XXX (XXX.X%) | |
| CS (Medical History) | XXX (XXX.X%) | |
| CS (Adverse Event) | XXX (XXX.X%) | |

#### 14.3.7 Vital Signs and Body Weight

- 14.3.7.1 Vital Signs Body Temperature [degree C]
- 14.3.7.2 Vital Signs Respiratory Rate [breaths/min]
- 14.3.7.3 Vital Signs Systolic Blood Pressure [mmHg]
- 14.3.7.4 Vital Signs Diastolic Blood Pressure [mmHg]
- 14.3.7.5 Vital Signs Heart/Pulse Rate [beats/min]
- 14.3.7.6 **Body Weight [kg]**

Use the layout <For continuous Laboratory Assessment>, clinical relevance {Normal, NCS, CS (Medical History), CS (Adverse Event)} analysis will be only presented for 14.3.7.1, 2, 3, 5.

Footnote "For Body Weight, uncheck of Clinical Relevance 'CS' will be recoded as 'Normal / NCS' for analysis".

Footnote "Baseline is Visit 2 (Day 1, Pre-dose) or alternatively as Visit 1 (Screening) if Visit 2 (Day 1, Pre-dose) data are not available".

Footnote for weight "Baseline is Visit 2 (Day 1) or alternatively as Visit 1 (Screening) if Visit 2 (Day 1) data are not available".



Careseng 1370 for Healthy Volunteers

#### 14.3.8 12-Lead Electrocardiogram (EKG)

#### 14.3.8.1 Electrocardiogram - Overall Interpretation

Population: Intent-to-Treat Population

| Characteristics | Dose Level |
|-------------------------------------------------------------|-------------|
| . (Adjusted) Visits, see visit table below 14.3 | |
| n (Missing) | XXX (XXX) |
| Normal | XXX (XX.X%) |
| NCS | XXX (XX.X%) |
| CS (Medical History) | XXX (XX.X%) |
| CS (Adverse Event) | XXX (XX.X%) |
| . Baseline to (Adjusted) Visits, see visit table below 14.3 | |
| n (Missing) | XXX (XXX) |
| Relieved | XXX (XX.X%) |
| Unchanged | XXX (XX.X%) |
| Worsened (Medical History) | XXX (XX.X%) |
| Worsened (Adverse Event) | XXX (XX.X%) |

- Baseline is Visit 2 (Day 1, Pre-dose) or alternatively as Visit 1 (Screening) if Visit 2 (Day 1, Pre-dose) data are not available.
- Refer to [Instructions and Abbreviations] of title pages for Transition of Clinical Relevance

#### 14.3.8.2 Electrocardiogram - Sinus Rhythm

Population: Intent-to-Treat Population

| Characteristics | Dose Level |
|--------------------------------------------------------|-------------|
| . (Adjusted) Visits, see visit table below 14.3 | |
| n (Missing) | XXX (XXX) |
| Normal | XXX (XX.X%) |
| Abnormal | XXX (XX.X%) |
| . Baseline to (Adjusted) Visits, see visit table below | v 14.3 |
| n (Missing) | XXX (XXX) |
| Normal to Abnormal | XXX (XX.X%) |
| No Change | XXX (XX.X%) |
| Abnormal to Normal | XXX (XX.X%) |

- Baseline is Visit 2 (Day 1, Pre-dose) or alternatively as Visit 1 (Screening) if Visit 2 (Day 1, Pre-dose) data are not available.
  - 14.3.8.3 Electrocardiogram Ventricular Rate [beats/min]
  - 14.3.8.4 Electrocardiogram PR Interval [msec]
  - 14.3.8.5 Electrocardiogram QRS Interval [msec]
  - 14.3.8.6 Electrocardiogram QT Interval [msec]
  - 14.3.8.7 Electrocardiogram QTc Interval [msec]

Use the layout <For continuous Laboratory Assessment>, excluding clinical relevance {Normal, NCS, CS (Medical History), CS (Adverse Event)} analysis

Footnote "Baseline is Visit 2 (Day 1, Pre-dose) or alternatively as Visit 1 (Screening) if Visit 2 (Day 1, Pre-dose) data are not available".



Version 1.0, 08-SEP-2022

**Protocol Number: Careseng 1370-01** 

A Phase I Dose-Escalation Study in Healthy Volunteers to Evaluate the Safety and Tolerability Profiles of Careseng 1370

Protocol version: 5.0, 18SEP2020

Sponsor:

Careseng 1370 for Healthy Volunteers

The Mock-up "Subject Data Listings" is planned according to ICH E3, in which relevant CSR section is 16.2. The words shadowed below are for notifications, or to be revised, or variables/format/footnotes to be included.

All listing will be sorted by (1) Eligibility {Eligible subjects by dose level, Screen failures} (2) Subject ID (3) Visit No. (4) Item No.

#### **Instructions and Abbreviations:**

(1) Subject ID contains Screening Number and Subject Number (SCSS-DRR) for eligible subject and Screening Number (SCSS) for non-eligible subject / screening failure.

| Site ID C | 1 = Taipei Medical University Hospital (TMUH) |
|---|---|
| Screening number SCSS | Assigned sequentially from SC01 for each site |
| Dose Level D | A = Careseng 1370 1 sachet before breakfast for consecutive 5 days B = Careseng 1370 1 sachet before breakfast and 1 sachet before lunch for consecutive 5 days C = Careseng 1370 1 sachet before breakfast and 2 sachets before lunch for consecutive 5 days |
| Subject Number DRR: | Assigned sequentially from $\boxed{D}01$ for dose level $\boxed{D}$ for each site |

#### (2) DP/AG:

D denotes dose level

- A: Careseng 1370 1 sachet before breakfast for consecutive 5 days
- B: Careseng 1370 1 sachet before breakfast and 1 sachet before lunch for consecutive 5 days
- C: Careseng 1370 1 sachet before breakfast and 2 sachets before lunch for consecutive 5 days
- D (1 sachet/day) (modified cohort): Careseng 1370 1 sachet before breakfast on 1st, 3rd and 5th days

#### P denotes population

I: intent-to-treat (ITT) population

- Volunteers receive any Careseng 1370

M: Maximum Tolerated Dose (MTD)-Evaluable Population, satisfying

- 1. A subset of ITT population
- 2. Experiences DLT OR with at least 80% of study drug compliance and has exposed to Careseng 1370 for at least 4 days

A denotes age in Y/O

Age = int((date of informed consent - date of birth)/365.25)

G denotes gender

M: male F: female

(3) Date format: YYYY-MM-DD

(4) For Visit Name (in Tables and Figures) and Visit Code (in Subject Data Listing):

| Visit No. | Visit Description | Visit Day | Visit Name | Visit Code |
|---|---|---|---|---|
| 1 | Visit 1 Screening Visit | <b>-14</b> ∼ <b>-1</b> | Visit 1 (Screening) | V01 |
| 2 | Visit 2 Hospitalization: Day -1 to Day 1 | 1 | Visit 2 (Day 1) | V02D01 |
| 3 | Visit 3 Discharge: Day 2 | 2 | Visit 3 (Day 2) | V03D02 |
| 4 | Visit 4: Day 3 | 3 | Visit 4 (Day 3) | V04D03 |
| 5 | Visit 5: Day 4 | 4 | Visit 5 (Day 4) | V05D04 |
| 6 | Visit 6 Hospitalization: Day 4 to Day 5 | 5 | Visit 6 (Day 5) | V06D05 |
| 7 | Visit 7 Discharge: Day 6 (24±2 hrs post-last dose) | 6 | Visit 7 (Day 6) | V07D06 |



Careseng 1370 for Healthy Volunteers

| Visit No. | Visit Description | Visit Day | Visit Name | Visit Code |
|---|---|---|---|---|
| 8 | Visit 8 Follow-up Visit: Day 7 | 7 | Visit 8 (Day 7) | V08D07 |
| 8 | (48±2 hrs post-last dose) | , | Visit o (Day 1) | V 00D07 |
| 9 | Visit 9 Follow-up Visit: Day 8 | 8 | Visit 9 (Day 8) | V09D08 |
| , | (72±2 hrs post-last dose) | | v isit / (Day 0) | V 09D00 |
| 10 | Visit 10 Follow-up Visit: Day 12±2 | 10 ~ 14 | Visit 10 (Day 12) | V10D12 |
| 1.1 | Visit 11 Final Visit | 22 | Visit 11 (Day 22) | V11D22 |
| 11 | (Day 22±2, within 3 days after withdrawal) | | | V11D22 |
| - | Unscheduled Visit | - | - | V□□.□ |

(5) For the visit/assessment days and hour (like AE Onset Day), they were derived by formula below Day/Hour = [visit/assessment date/time – the first treatment date/time + 1], if date/hour  $\geq 1^{st}$  dosing date/time,

Day/Hour = [visit/assessment date/time – the first treatment date/time], if date/hour < 1<sup>st</sup> dosing date/time, Duration in days/hours = [end date/time – onset date/time + 1] if end date/time is active

Duration in days/hours = [end date/time – onset date/time] if end date/time is inactive

(6) Full term for 'Protocol Deviation Code':

| Code | Full Term |
|---|---|
| | <to added="" be="" data="" final="" in="" real="" tabulation="" upon=""></to> |

#### (7) Full term for Laboratory Measurements:

#### Hematology

| Test code of SDTM | Test of SDTM | Test in section 14 |
|---|---|---|
| HGB | Hemoglobin | Hemoglobin |
| HCT | Hematocrit | Hematocrit (Hct) |
| RBC | Erythrocytes | RBC |
| WBC | Leukocytes | WBC |
| NEUTLE | Neutrophils/Leukocytes | Neutrophils |
| LYMLE | Lymphocytes/Leukocytes | Lymphocytes |
| MONOLE | Monocytes/Leukocytes | Monocytes |
| EOSLE | Eosinophils/Leukocytes | Eosinophils |
| BASOLE | Basophils/Leukocytes | Basophils |
| NEUT | Neutrophils | Absolute neutrophil Count (ANC) |
| LYM | Lymphocytes | Lymphocyte Count |
| PLAT | Platelets | Platelet |
| INR | Prothrombin Intl. | International normalized ratio (INID) |
| INK | Normalized Ratio | International normalized ratio (INR) |
| ACTIVATED Partial | | Activated partial thromboplastin |
| APTT | Thromboplastin Time | time (APTT) |

#### Biochemistry

| Test code of SDTM | Test of SDTM | Test in section 14 |
|---|---|---|
| AST | Aspartate Aminotransferase | AST, SGOT |
| ALT | Alanine Aminotransferase | ALT, SGPT |
| ALB | Albumin | Albumin |
| ALP | Alkaline Phosphatase | Alkaline Phosphatase (ALP) |
| BILI | Bilirubin | Total bilirubin |
| CREAT | Creatinine | Creatinine |
| UREAN | Urea Nitrogen | Blood urea nitrogen (BUN) |
| CRP | C Reactive Protein | C-reaction protein (CRP) |
| PROT | Protein | Total protein |
| GGT | Gamma Glutamyl Transferase | Gamma-glutamyl transferase ( $\gamma$ - |
| | | GT) |



Careseng 1370 for Healthy Volunteers

| Test code of SDTM | Test of SDTM | Test in section 14 |
|-------------------|---------------|--------------------|
| GLUC | Glucose | Blood Glucose |
| URATE | Urate | Uric Acid |
| CHOL | Cholesterol | Total Cholesterol |
| TRIG | Triglycerides | Triglyceride (TG) |
| SODIUM | Sodium | Sodium (Na) |
| K | Potassium | Potassium (K) |
| CA | Calcium | Calcium (Ca) |
| MG | Magnesium | Magnesium |
| PHOS | Phosphate | Phosphorus |
| AMYLASE | Amylase | Amylase |
| LIPASET | Lipase | Lipase |

#### Urinalysis

| Of Mary 313 | | |
|-------------------|--------------|--------------------|
| Test code of SDTM | Test of SDTM | Test in section 14 |
| PH | pН | pH |
| PROT | Protein | Protein |
| RBC | Erythrocytes | RBC |
| WBC | Leukocytes | WBC |
| CASTS | Casts | Casts |

#### • Immunology

| Test code of SDTM | Test of SDTM | Test in section 14 |
|-------------------|---------------|--------------------|
| CD3 | CD3+ | CD3+ |
| CD3CD4 | CD3+/CD4+ | CD3+/CD4+ |
| CD3CD8 | CD3+/CD8+ | CD3+/CD8+ |
| CD19 | CD19+ | CD19+ |
| CD16CD56 | CD16+/CD56+ | CD16+/CD56+ |
| CD4CD8 | CD4/CD8 Ratio | CD4/CD8 Ratio |

#### (8) For Serial No.,

- HXXX: Serial No. of General Medical History,
- $C|\overline{X}|\overline{X}|\overline{X}|$ : Serial No. of Concomitant Medication
- AXXX: Serial No. of Adverse Event
- COXX: Serial No. of Comment

#### (9) For clinical relevance,

- NCS denotes 'abnormal but not clinically significant'
- CS denotes 'abnormal and clinically significant'

#### (10) General abbreviations

| Code | Full Term |
|------------|------------------------|
| A, NA, N/A | Not Applicable |
| U, UK, U/K | Unknown |
| O, OG, O/G | Ongoing |
| D, ND, N/D | Not Done |
| M, MS, M/S | Missing |
| MH | Medical History |
| AE | Adverse Event |
| CM | Concomitant Medication |
| INCXX | Inclusion Criterion XX |
| EXCXX | Exclusion Criterion XX |

Careseng 1370 for Healthy Volunteers

#### 16.2 Subject Data Listings

### 16.2.1 Discontinued Subjects

16.2.1.1 Screen Failures

Screening failure reasons and criteria (IE)

16.2.1.2 Study Termination of Eligible Subjects

First Treatment Date/Day,

Last Treatment Date/Day,

Study Termination Date, Study Duration [days] (Refer to table 14.1.2 for formula),

Status (Study Completed or Not Completed),

Primary Discontinued Reason and Description.

16.2.1.3 Visit Dates and Inform Consent Date

Including visit status and fasting status

16.2.1.4 Visit Adjustment

(If any)

16.2.1.5 Unscheduled Visit Dates

(If any)

16.2.1.6 Protocol Versions Applied

#### 16.2.2 Protocol Deviations

16.2.2.1 Inclusion / Exclusion Criteria

Including visit and protocol version if there is related protocol amendment.

16.2.2.2 Protocol Deviations

Including Subject ID / Severity / Code / Description / Population to be excluded,

† according to ICH E9 section '5.2.2 Per Protocol Set', protocol violations may include errors in treatment assignment, the use of excluded medication, poor compliance, loss to follow-up and missing data.

16.2.2.3 Non Protocol Deviation Findings

#### 16.2.3 Eligible Subjects Excluded from the Safety/Efficacy Analysis

- 16.2.3.1 Eligible Subjects Excluded from ITT Population
- 16.2.3.2 Eligible Subjects Excluded from MTD-Evaluable Population

#### 16.2.4 Demographic Data and Baseline Characteristics

16.2.4.1 Demographic Data

Including re-screen status, preceding Screening No., body height, baseline weight and BMI

16.2.4.2 General Medical History

Identifier of current condition included

Footnote: Current condition lists the medical histories that are ongoing or with end date > date of visit 1

16.2.4.3 Chest X-ray



Careseng 1370 for Healthy Volunteers

# 16.2.5 Concomitant Medications, Treatments, Procedures and Prohibited Foods

- 16.2.5.1 Medication History & Concomitant Medications
- 16.2.5.2 Prohibited Foods

#### 16.2.6 Study Drug Administration, Compliance and Exposure

- 16.2.6.1 Study Drug Compliance and Exposure
  Including Total IP Administration [Sachets], Treatment Duration [Days], Treatment
  Compliance [%], Mean Daily Dose [Sachet / day]
  Refer to table 14.1.6 for the definition
- 16.2.6.2 Drug Accountability

#### 16.2.7 Adverse Event (AE) and Serious Adverse Event (SAE)

- 16.2.7.1 Pre-Treatment AE
- 16.2.7.2 Treatment Emergent AE

Variables: In addition to event description and general AE profiles (Before / After doseing, onset date, resolution date, severity, relationship to study treatment, action taken to study treatment, seriousness, outcome), the Subject data listing will also present the MedDRA System Organ Class and preferred term, onset day, and AE duration [days]

#### Footnote:

- Onset Day = onset date the first treatment dosing date + 1
- AE duration [days]
  - = resolution date onset date (while resolved)

=study exit date - onset date (while not resolved, noted with '+')

- 16.2.7.3 Treatment Emergent AE Treatment Related AE

  Treatment Related is defined as Definitely Related, Probable Related, or Possibly Related
- 16.2.7.4 Treatment Emergent AE DLT
- 16.2.7.5 Treatment Emergent AE − Grade ≥3 AE
- 16.2.7.6 Treatment Emergent AE − Grade ≥3 Treatment Related AE
- 16.2.7.7 Treatment Emergent AE AE Leading to Action Taken
- 16.2.7.8 Serious Adverse Event (SAE)
- 16.2.7.9 Suspected Unexpected Serious Adverse Reaction (SUSAR) (Unexpected Treatment Related SAE)

#### **16.2.8** Laboratory Examination

- 16.2.8.1 Laboratory Examination Summary in Standard Unit
- 16.2.8.2 Laboratory Examination Hematology
- 16.2.8.3 Laboratory Examination Biochemistry
- 16.2.8.4 Laboratory Examination Urinalysis
- 16.2.8.5 Laboratory Examination Immunology
- 16.2.8.6 Laboratory Examination Not Done Reason and Comments



Careseng 1370 for Healthy Volunteers

16.2.8.7 Pregnancy Test For Female Subjects Only

#### **16.2.9** Other Safety Measurements

- 16.2.9.1 Physical Examination
- 16.2.9.2 Physical Abnormalities
- 16.2.9.3 Vital Signs and Body Weight
- 16.2.9.4 12-Lead Electrocardiogram (EKG)

Variables: Overall interpretation, Sinus Rhythm, Ventricular Rate, PR Interval, QRS Interval, QT Interval, QTc Interval

16.2.9.5 Not Done Reason and Comments of Other Safety Measurements

### 16.2.10 Pharmacokinetics Sampling

PK blood sampling time points:

| 1 | it blood sampling | time points. | |
|---|-------------------|-----------------|------------|
| ſ | V02D01 Pre-Dose | V06D05 Pre-Dose | V07D06 24h |
| | V03D02 Pre-Dose | V06D05 0.5h | V08D07 48h |
| | V04D03 Pre-Dose | V06D05 1h | V09D08 72h |
| | V05D04 Pre-Dose | V06D05 2h | |
| | | V06D05 4h | |
| | | V06D05 6h | |
| | | V06D05 12h | |

16.2.10.1 Blood Sampling Time

#### **16.2.11** Comments

16.2.11.1 Comment

Version 1.0, 08-SEP-2022 Protocol No.: Careseng 1370-01